CLINICAL TRIAL: NCT04008264
Title: A Novel Usage of Transdermal Scopolamine in Reducing Narcotic Usage in Outpatient Hand Surgery
Status: Completed | Type: Observational
Sponsor: Alexander M Spiess, MD (Other)
Responsible Party: Sponsor-Investigator, Alexander M Spiess, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY18100076
Record Dates: First submitted 2019-06-20; First posted 2019-07-05 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Post Operative Pain Management
MeSH Terms: interventions — Butylscopolammonium Bromide; Scopolamine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard post operative pain regimen: There will be a 3 month pre-intervention phase where participants will be placed on a standard post-operative analgesic regimen consisting of an opioid, a NSAID, and acetaminophen. Patients will record their narcotic and non-opioid analgesic usage patterns in the two weeks following outpatient hand surgery.
- Scopolomine group: During the observational phase, patients will be on scopolamine for a total 6 day course (one patch applied at time of surgery, prescription for one patch), and patients will record their narcotic and non-opioid analgesic usage patterns in the two weeks following outpatient hand surgery. The patients who incorporate scopolamine into their post operative analgesia regimen will be eligible for inclusion in the study.
  Interventions: Drug: Scopolamine Patch (Transderm V)

INTERVENTIONS:
Drug: Scopolamine Patch (Transderm V) — During the observational phase, patients will be given a prescription for an 18 day supply of scopolamine, and patients will record the same data as prior to the intervention.
  Other Names: Transderm Scop
  Groups: Scopolomine group

SUMMARY:
The investigators will examine and analyze opioid narcotic usage patterns by requesting patients keep a two week log of their opioid usage following outpatient hand surgery with a standard analgesic regimen consisting of an opioid, NSAID, and acetaminophen. Following a pre-intervention period, the investigators will add scopolamine to the regimen and have patients monitor their opioid consumption. The investigators will then compare opioid consumption patterns following completion of the study.

DETAILED DESCRIPTION:
Aim 1: Determine whether the addition of transdermal scopolamine to a standard analgesic regimen reduces opioid utilization following outpatient hand surgery as reported by patients Objectives: The investigators will compare opioid usage between patients who complete logs during the pre-intervention stage of the study and the intervention stage of the study to determine the effect of including scopolamine as a medication in standard post-operative analgesic regimens following outpatient hand surgery. As this is the primary objective of our study, an a priori power analysis was conducted. Based on a two-sided two-sample independent t-test with a specified significant level of 0.05, a power of 0.8, and a moderate effect size of 0.5; 64 patients will need to complete each portion of the study to provide an overall sample size of 128 patients.

Outcome Variables and Analysis: The absolute number of logged opioid use during the two-week study period will be compared between the pre-intervention and intervention groups using a two-sided independent samples t-test.

Aim 2: Determine patient compliance with usage of multi-modal analgesic medications and the feasibility of supplementing with an additional agent Objectives: During the pre-intervention stage of the trial, the investigators will encourage patients to utilize non-opioid analgesics over opioids and have patients keep a log of their NSAID and acetaminophen usage. This aim will partially establish whether patients are being adequately counseled regarding multi-modal pain control as patients with high opioid consumption should also have high rates of use of their non-opioid analgesics. It will also establish whether it is feasible to expect patients to comply with the introduction of novel medications into analgesic regimens. It will establish baseline rates of non-narcotic pain medication use overall and stratified by procedure. It may also further support the existing evidence that non-opioid pain medications reduce opioid requirements while providing more significant pain relief than opioids alone.

Outcome Variables and Analysis: Data analyzed will include percentage of individual non-opioid pain medications used (prescriptions will be provided so patient could take medication around the clock), patient pain scores, and percentage of opioids used. Percentages of non-opioid pain medications and opioid pain medications will be compared on a patient-by-patient basis by utilizing a paired t-test. The association between patient perceived pain levels and percentage of each medication used will be determined with multiple linear regression.

Aim 3: Aim 3: Assess patient and operative factors that contribute to prolonged or greater than expected opioid usage.

Objectives: The factors contributing to prolonged patient use of opioids and need for repeated refills are poorly understood. An analysis of factors contributing to prolonged opioid use and a determination of baseline opioid use rates would allow hand surgeons to have a better understanding of factors that may place a patient at risk or to identify when patients are exceeding the typical requirements for opioids. Identification of these patients may allow for increased counseling, referral to a pain specialist, or increased surveillance. Details of the operative procedure and typical narcotic requirements will guide providers in prescribing more limited opioid prescriptions appropriate to an individual procedure with few to no refills authorized.

Outcome Variables and Analysis: Patients will be separated into groups based on whether they used over 80% of their opioid prescription or if they requested a refill of their opioid prescription within the two week study period. A univariate analysis of patient demographic factors and operative details will identify factors that are potentially associated with higher rates of opioid consumption following surgery. Chi square tests will be performed for categorical variables and student's t-tests will be used for continuous variables. Binary logistic regression will then be performed using variables identified in the univariate screen in order to identify independent factors contributing to a higher number of opioids used after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-55 undergoing outpatient hand and wrist surgery via sedation and a regional block
* Procedures eligible for inclusion will be limited to those involving the wrist and the hand.

Exclusion Criteria:

* Patients undergoing procedures under local, regional anesthesia alone, sedation alone, and general endotracheal anesthesia
* Patients with a history of acute angle closure or open angle glaucoma;
* History of drug hypersensitivity to scopolamine, other belladonna alkaloids, or any other ingredient or component in the formulation or delivery system;
* History of previous gastrointestinal or urinary bladder obstruction;
* History of seizures or psychosis; patients with hepatic or renal impairment;
* Patients under the age of 18 or over the age of 55;
* Patients who are currently pregnant or nursing.
* Patients currently using prescription opioids for other chronic medical conditions or who are actively using heroin.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Patients between the ages of 18-55 undergoing outpatient hand and wrist surgery via sedation and a regional block
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of opioids taken during study period | 21 days
  Determine whether the addition of transdermal scopolamine to a standard analgesic regimen reduces opioid utilization following outpatient hand surgery as reported by patients. The outcomes will be measured through review of post operative pain medication logs, and outcome surveys.

SECONDARY OUTCOMES:
Number of non-opioid analgesics taken during study period | 21 days
  Determine patient compliance with usage of multi-modal analgesic medications and the feasibility of supplementing with an additional agent.The outcomes will be measured through review of post operative pain medication logs, and outcome surveys. Will record number of doses taken of tylenol and ibuprofen

OTHER OUTCOMES:
Pain Medication Usage beyond 20 day study period | 9 months
  Assess patient and operative factors that contribute to prolonged or greater than expected opioid usage. The outcomes will be measured through review of post operative pain medication logs, and outcome surveys. The patient and operative factors and will be determined from review of the chart and personal interview of the patient. Patients who continue to take pain medications beyond 20 days will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Spiess, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Falk Clinic, 3601 Fifth Ave., Suite 6B, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT04008264/Prot_SAP_001.pdf